CLINICAL TRIAL: NCT04908956
Title: A Multicentre Single-arm Phase II Trial Assessing the Safety and Efficacy of First-line Osimertinib and Locally Ablative Radiotherapy in Patients With Synchronous Oligo-metastatic EGFR-mutant Non-small Cell Lung Cancer
Brief Title: Osimertinib and Locally Ablative Radiotherapy in Patients With Synchronous Oligo-metastatic EGFR Mutant NSCLC (STEREO)
Acronym: STEREO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial struggled with low activation due to the COVID pandemic. The Steering Committee took the decision to close the accrual in the STEREO trial as of 31 October 2023. It is important to note that no safety concerns have led to this decision.
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 17-20; 2020-004114-35 (EudraCT Number); ESR-19-20384 (Other: AstraZeneca)
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: NSCLC Stage IV; EGFR Gene Mutation
Keywords: NSCLC; EGFR mutation (exon 19 deletion and/or exon 21 L858R); Osimertinib; SBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib & SBRT (Experimental): Osimertinib 80mg once daily p.o., until progression or unacceptable toxicity & locally ablative radiotherapy (SBRT) to the primary tumour and to all metastatic sites.
  Interventions: Drug: Osimertinib; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Osimertinib — Osimertinib is a Tyrosine Kinase Inhibitor (TKI). It is an irreversible inhibitor of Epidermal Growth Factor Receptors (EGFRs) harboring sensitising-mutations (EGFRm) and TKI-resistance mutation T790M.
  The appropriate number of osimertinib tablets (80 mg or 40 mg if the dose is reduced due to toxicity) will be provided to patients to be self-administered at home.
  Other Names: Tagrisso
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered using risk-adapted SBRT with a maximum of 5 SBRT fractions.

SUMMARY:
STEREO is single-arm phase II study, which aims to evaluate the safety and efficacy of osimertinib combined with early locally ablative radiotherapy of all cancer sites in patients with synchronous oligo-metastatic (primary tumour and maximum 5 metastases) EGFR-mutant (exon 19 deletion or exon 21 L858R) NSCLC. Eradication of all macroscopic cancer sites at the time of primary diagnosis by combined modality treatment is expected to decrease the risk of resistance development with only microscopic disease potentially remaining. This will result in an improvement of PFS and OS without added high-grade toxicity.

DETAILED DESCRIPTION:
Targeting Epidermal Growth Factor Receptor (EGFR) mutation has fundamentally changed the treatment of metastatic Non-Small Cell Lung Carcinoma (NSCLC).

Several randomised phase III studies have compared first-generation (erlotinib or gefitinib) or second-generation (afatinib) EGFR-targeting TKIs with standard platinum-based chemotherapy and all reported significantly improved objective response rates (ORR) and progression-free survival (PFS). For patients with TKI resistance development by T790M mutation, which is the resistance mechanism in about 50% of the patients, osimertinib is superior compared to platinum-based chemotherapy with significant and clinically relevant improved ORR and PFS. Recently, the FLAURA study reported improved PFS of osimertinib compared to first-generation TKI (erlotinib or gefitinib) for untreated EGFRmutant advanced NSCLC, without differences in ORR. On longer follow-up, first-line osimertinib was also associated with improved survival.

Integration of local therapy into a multimodality treatment is a promising strategy to overcome the limitations of EGFR-targeting TKIs alone, despite patients suffering from a metastatic stage of disease. This is based on the observations that disease progression under EGFR-targeting TKI most frequently occurs at the original sites of metastatic disease and that the majority of patients show disease progression in a limited number of metastatic lesions, a situation defined as oligoprogression. Al-Halabi et al. reported in a series of 49 patients that 47.0%, 32.6%, and 20.4% of the patients developed original site failure, combined original site and distant site failure and distant site failure as first progression of disease to EGFR-targeting TKI. Primary tumour size was the most significant predictor for original site failure. Li et al. reported about 266 patients treated with first-line EGFR-targeting TKI and disease progression was reported at original and distant sites in 39% and 61%, respectively. Guo et al. reported disease progression in original sites, combined original and distant sites and distant sites in 50%, 28% and 22%, respectively. Consequently, EGFR-targeting TKIs appear less effective in controlling sites of macroscopic disease, where residual cancer cells ultimately acquire resistance and become the source of further disease progression.

Early imaging-based detection of oligoprogressive disease sites and their local ablation combined with continuation of TKI is one strategy to overcome this resistance development: metastatic sites with acquired resistance to EGFR-targeting TKI are eradicated by locally ablative treatment, irrespective of the underlying resistance mechanism, whereas non-progressing and EGFR-sensitive sites are continuously targeted and controlled by TKI therapy. This combined modality strategy has shown promising results in several retrospective studies, including a recent Swiss cohort study, where locally ablative treatment added to continuation of osimertinib in oligoprogressive T790M-mutant NSCLC patients was identified as the intervention which prolonged overall survival (OS). A randomised phase II trial is currently testing this hypothesis of locally ablative radiotherapy for oligoprogressive driver mutated NSCLC patients (NCT03256981); assessment of liquid biopsy for response evaluation is an important translational endpoint to identify patients with residual resistant disease after locally ablative treatment.

However, the strategy of local eradication of oligoprogressive disease has the limitation that imaging can only detect resistance development when this has already translated into macroscopically progressive disease. Systemic dissemination of resistant disease beyond the initial sites of acquired resistance development may then have already occurred, which is supported by the finding that the majority of patients develop further disease progression after locally ablative treatment. Consequently, there is a strong rationale of early targeting of local disease sites at high risk for developing acquired EGFR resistance, before imaging-based progression has developed. This strategy is supported by retrospective data of patients with brain metastases, where early radiosurgery combined with EGFR-targeting TKI improved OS compared to EGFR-targeting TKI alone and delayed radiotherapy at the time of disease progression (HR 0.39, 46 months vs 25 months). The hypothesis of upfront SBRT is supported by a recent randomised phase III trial of patients with oligo-metastatic EGFR-mutated NSCLC treated with first-generation EGFR TKIs presented at ASCO 2020, which demonstrated a PFS and OS benefit for early use of SBRT compared to systemic therapy alone. However, this study is limited by the use of first-generation TKIs only, and especially by chemotherapy as mandatory second line treatment.

The value of combined modality systemic therapy with locally ablative therapy for oligo-metastatic NSCLC has recently been evaluated in several randomised trials. All studies reported a significantly and clinically relevant improved OS or PFS for adding locally ablative therapy to standard of care systemic therapy. However, these studies included only very few NSCLC patients with activating driver mutations and the benefit of adding upfront local radiotherapy might be smaller or larger in this NSCLC patient population with activating driver mutations and treatment with TKIs: smaller because of the higher systemic efficacy of TKIs compared to chemotherapy or larger because the benefit of local treatment might become most obvious if potential microscopic disease is successfully controlled by TKIs.

Consequently, there is a clinical need to evaluate locally ablative therapy in oligo-metastatic EGFR-mutant NSCLC patients and simultaneously a strong rationale that this population might benefit in particular from a combined modality treatment: the benefit of locally ablative therapy is expected to be largest in situations of effective systemic therapies to control locally untreated microscopic disease which is true for EGFR targeting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, treatment naïve EGFR-mutant NSCLC, with or without T790M resistance mutation. Presence of the sensitising EGFR-mutation (exon 19 deletion and/or exon 21 L858R) detected by an accredited laboratory.
* Synchronous oligo-metastatic stage IV disease (max 5 lesions)
* Measurable disease as defined according to RECIST v1.1
* All lesions amenable for radical radiotherapy according to local judgment
* Age ≥18 years
* ECOG performance status 0-2
* Life expectancy ≥12 months
* Adequate haematological, renal & liver function
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 7 days before enrolment.
* Written IC for protocol treatment

Exclusion Criteria:

* Prior chemotherapy, immunotherapy, radiotherapy or therapeutical surgery for NSCLC (an exception is the resection and postoperative radiotherapy of the resection cavity of CNS or adrenal metastases)
* More than 5 distant oligo-metastases (any second intra-thoracic lesion will count as a distant metastasis; regional nodal metastases will not count towards 5 oligo-metastases) and more than 2 intra-thoracic lesions.
* Brain metastases not amenable for radiosurgery or neurosurgery
* Presence of leptomeningeal metastases
* Symptomatic spinal cord compression
* Extracranial metastatic locations not amenable for radical radiotherapy
* Currently receiving medications or herbal supplements known to be potent CYP3A4 inducers
* Any evidence of severe or uncontrolled systemic diseases
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* Any of the following cardiac criteria: QTcF >470 msec; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG; Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
* Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
* Idiopathic pulmonary fibrosis which is a contraindication to lung radiation.
* History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial and up to 6 weeks for women and up to 4 months for men, after the last osimertinib dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Safety of first-line EGFR-targeting osimertinib and SBRT to the primary tumour and all metastases | Rate of grade ≥2 pneumonitis, requiring medical treatment, any time during the first 18 months on trial follow-up
  Defined as the number of patients experiencing grade ≥2 pneumonitis, requiring medical treatment, any time during the first 18 months post enrolment over the total number of patients in the primary-endpoint safety cohort.
Efficacy of first-line EGFR-targeting osimertinib and SBRT to the primary tumour and all metastases | Time from the date of enrolment until documented progression or death, if progression is not documented, assessed for a maximum of approx. 44 months after enrolment of the first patient
  If safety is proven, efficacy will be hierarchically tested in terms of Progression-free survival (PFS) according to RECIST v1.1, in the efficacy cohort.
  PFS is defined as the time from the date of enrolment until documented progression or death, if progression is not documented.

SECONDARY OUTCOMES:
Overall survival (OS) | Time from the date of enrolment until death from any cause. Censoring will occur at the last follow-up date, assessed for a maximum of approx. 44 months after enrolment of the first patient
  Defined as the time from the date of enrolment until death from any cause.
Pattern of disease progression | Evaluated up to 18-months post enrolment
  Defined as the pattern of disease progression is defined as the site of first progression: None, locoregional, distant (bone, brain, liver, etc.) or both locoregional and distant
Distant progression-free survival | Time from date of enrolment until development of new metastases, excluding oligo-metastases diagnosed at enrolment - assessed for a maximum of approx. 44 months after enrolment of the first patient
  Defined as the time from date of enrolment until development of new metastases, excluding oligo-metastases diagnosed at enrolment
Objective response rate | Time from enrolment across all trial assessment time-points - assessed for a maximum of approx. 44 months after enrolment of the first patient
  Defined as the percentage of patients that achieve a best overall response [complete response (CR) or partial response (PR)] according to RECIST v1.1
Duration of response | From the date of first documentation of objective response to the date of first documented progression, relapse or death- assessed for a maximum of approx. 44 months after enrolment of the first patient
  Defined as the interval from the date of first documentation of objective response (CR or PR, according to RECIST v1.1) to the date of first documented progression, relapse or death
Adverse events according to CTCAE v5.0 | Assessed for a maximum of approx. 44 months after enrolment of the first patient
  To assess the safety and tolerability of the treatment.
Symptom-specific and global quality of life | Assessed from baseline to 24 weeks on treatment
  QoL will be assessed by the Lung Cancer Symptom Scale, a 9-item questionnaire including six symptoms (i.e., appetite loss, fatigue, cough, dyspnoea, haemoptysis and pain) and three items addressing symptomatic distress, normal activity, and global QoL. The primary QoL endpoints will be the change in the LCSS total score (average of all 9 items) from baseline to 24 weeks on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, MD-PhD, Study Chair — University Hospital, Zürich
Locations (18):
- Italy (3):
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - Instituto Europeo di Oncologia (IEO), Milan
  - AULSS2 Marca Trevigiana Treviso, Treviso
- Netherlands (2):
  - The Netherlands Cancer Institute Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
- Medical University Gdansk, Gdansk, Poland
- National University Hospital, Singapore, Singapore
- South Korea (2):
  - National Cancer Center, Goyang-si
  - Severance Hospital, Yonsei University Health System, Sinchŏn-dong
- Spain (5):
  - Hospital General de Alicante, Alicante
  - Vall d'Hebron University Hospital, Barcelona
  - Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona
  - Centro Integral Oncologíco Clara Campal (CIOCC) HM Hospitales, Madrid
  - Hospital Clínico de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Zürich USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Background] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Background] Weickhardt AJ, Scheier B, Burke JM, Gan G, Lu X, Bunn PA Jr, Aisner DL, Gaspar LE, Kavanagh BD, Doebele RC, Camidge DR. Local ablative therapy of oligoprogressive disease prolongs disease control by tyrosine kinase inhibitors in oncogene-addicted non-small-cell lung cancer. J Thorac Oncol. 2012 Dec;7(12):1807-1814. doi: 10.1097/JTO.0b013e3182745948. PMID 23154552
- [Background] Wang X, Zeng M. First-line tyrosine kinase inhibitor with or without aggressive upfront local radiation therapy in patients with EGFRm oligometastatic non-small cell lung cancer: Interim results of a randomized phase III, open-label clinical trial (SINDAS) (NCT02893332). Journal of Clinical Oncology 2020; 38(15_suppl): 9508-
- [Background] Misale S, Fatherree JP, Cortez E, Li C, Bilton S, Timonina D, Myers DT, Lee D, Gomez-Caraballo M, Greenberg M, Nangia V, Greninger P, Egan RK, McClanaghan J, Stein GT, Murchie E, Zarrinkar PP, Janes MR, Li LS, Liu Y, Hata AN, Benes CH. KRAS G12C NSCLC Models Are Sensitive to Direct Targeting of KRAS in Combination with PI3K Inhibition. Clin Cancer Res. 2019 Jan 15;25(2):796-807. doi: 10.1158/1078-0432.CCR-18-0368. Epub 2018 Oct 16. PMID 30327306
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Background] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074